CLINICAL TRIAL: NCT05230680
Title: Multicenter, Open Label, Phase I/II of Azacitidine-CHOP for Patients With Nodal T-cell Lymphoma With T-follicular Helper Phenotype
Brief Title: Azacitidine-CHOP for Patients With Nodal T-cell Lymphoma With T-follicular Helper Phenotype (ACANTUS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Won Seog Kim (Other)
Responsible Party: Sponsor-Investigator, Won Seog Kim, Principal Investigator, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09-142
Record Dates: First submitted 2022-01-11; First posted 2022-02-09 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm ACHOP (Experimental): 1. Phase I Azacitidine D1-3 + CHOP (Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone)
     * Level 1 - Azacitidine 50mg/m2 D-2, -1, 1
     * Level 2 - Azacitidine 75mg/m2 D-2, -1, 1
     * Level 3 - Azacitidine 100mg/m2 D-2, -1, 1
     * Level 4 - Azacitidine 125mg/m2 D-2, -1, 1
  2. Phase II
     * Azacitidine D-2, -1, 1 + CHOP(Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone)
     * 6 cycles in total
  Interventions: Drug: ACHOP

INTERVENTIONS:
Drug: ACHOP — 1. Phase I Azacitidine D-2~D1, starting from dose level 1. Based on the BOIN design described above, if no DLT is identified in level 1, the dose will be escalated stepwise to levels 2, 3, and then 4.
     Azacitidine combined with CHOP regimen every 3 weeks as below:
     * Level 1 - Azacitidine 50mg/m2 D-2, -1, 1
     * Level 2 - Azacitidine 75mg/m2 D-2, -1, 1
     * Level 3 - Azacitidine 100mg/m2 D-2, -1, 1
     * Level 4 - Azacitidine 125mg/m2 D-2, -1, 1
     Azacitidine at each level will be combined with the corresponding CHOP regimen as follows:
     * Cyclophosphamide 750mg/m2 d1
     * Doxorubicin 50 mg/m2 d1
     * Vincristine 1.4 mg/m2 (Max: 2 mg) d1
     * Prednisolone 100mg PO d1-5
  2. Phase II
     * Azacitidine determined dose daily for D-2, -1, 1
     * CHOP (Cyclophosphamide 750mg/m2 d1, Doxorubicin 50 mg/m2 d1, Vincristine 1.4 mg/m2 (Max: 2 mg) d1, Prednisolone 100mg PO d1-5), 6 cycles in total

SUMMARY:
Induction treatment (every 3 weeks, total 6 cycles)

* Azacitidine D-2, -1, 1 (level 1: 50mg/m2, level 2: 75mg/m2, level 3: 100mg/m2, level 4: 125mg/m2)
* Cyclophosphamide 750mg/m2 d1
* Doxorubicin 50 mg/m2 d1
* Vincristine 1.4 mg/m2 (Max: 2 mg) d1
* Prednisolone 100mg PO d1-5 Maintenance treatment (every 4 weeks, total 12 cycles)
* Azacitidine 75mg/m2 d1-5

DETAILED DESCRIPTION:
1. Phase I Azacitidine will be administered intravenously from d-2 to d1, starting from dose level 1. Based on the BOIN design described above, if no DLT is identified in level 1, the dose will be escalated stepwise to levels 2, 3, and then 4.

   Subjects will receive intravenous azacitidine combined with CHOP regimen every 3 weeks as below:

   Level 1 - Azacitidine 50mg/m2 D-2, -1, 1 Level 2 - Azacitidine 75mg/m2 D-2, -1, 1 Level 3 - Azacitidine 100mg/m2 D-2, -1, 1 Level 4 - Azacitidine 125mg/m2 D-2, -1, 1

   Azacitidine at each level will be combined with the corresponding CHOP regimen as follows:
   * Cyclophosphamide 750mg/m2 d1
   * Doxorubicin 50 mg/m2 d1
   * Vincristine 1.4 mg/m2 (Max: 2 mg) d1
   * Prednisolone 100mg PO d1-5
2. Phase II

   * Azacitidine determined dose daily for D-2, -1, 1, Cyclophosphamide 750mg/m2 d1, Doxorubicin 50 mg/m2 d1, Vincristine 1.4 mg/m2 (Max: 2 mg) d1, Prednisolone 100mg PO d1-5 (6 cycles in total)
   * Use prophylactic trimethoprim-sulfamethoxazole 1T from the day of study drug administration to 21 days after the last dose of study treatment
   * Administer Peg-GCSF on study d2.
   * After Cycle 2, the study treatment can be administered if the ANC has been restored to ≥1,500/μL and platelets to ≥75,000/μL, and non-hematological toxicities that occurred in the previous cycle, except alopecia, have resolved to Grade 1 or less on d1 of each cycle.
   * If these hematological and non-hematological toxicities are not resolved, the clinical trial can be delayed for up to 21 days.
3. Consolidation therapy

   * After completing the planned first-line therapy in the clinical trial, the following consolidation therapy should be performed, regardless of the azacitidine dose level.
   * Azacitidine 75mg/m2 d1-5 (every 4 weeks, total 12 cycles)

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-naïve patients with newly diagnosed nodal T-cell lymphoma with T-follicular helper (TFH) phenotype as determined by the following 2016 WHO diagnostic criteria:

   * Angioimmunoblastic T-cell lymphoma
   * Follicular helper T-cell lymphoma
   * Peripheral T-cell lymphoma with follicular helper T-cell type
2. 20 to 85 years of age at diagnosis
3. ECOG performance status 0-2
4. Cardiac function suitable for chemotherapy: LVEF ≥45% on echocardiography or MUGA
5. Appropriate renal function: Serum Cr ≤2.0mg/dL or eGFR ≥ 30mL/min according to the Cockroft-Gault formula
6. Appropriate hepatic function: ALT ≤2.5x upper limit of normal (ULN) (or ≤5x ULN in the presence of liver involvement), total bilirubin ≤2x ULN (or ≤3x ULN in the presence of liver involvement)
7. Appropriate hematologic findings: absolute neutrophil count (ANC) ≥1,500/μL, platelets ≥100,000/μL (or ANC ≥500/μL and platelets ≥50,000/ μL in the presence of bone marrow involvement)
8. Written informed consent to participate in the study
9. Capable of following the study visit schedule and other requirements in the protocol
10. For women of childbearing potential, a negative pregnancy test
11. Women of childbearing potential must use an effective method of contraception (i.e., hormonal contraception, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) during the study period and for 3 months afterward. Men are to use an effective method of contraception during the study period and for 3 months afterward.
12. Life expectancy ≥90 days (3 months)
13. Hepatitis B or C infection: Hepatitis B carriers and subjects with inactive hepatitis C infection (normal levels of aminotransferases) are eligible if they take prophylactic antiviral drugs

Exclusion Criteria:

1. Other subtypes of non-Hodgkin's lymphoma
2. History of chemotherapy for Hodgkin's or other non-Hodgkin's lymphoma in the last 5 years
3. History of active cancer diagnosed within the last 3 years (with the exception of completely resected non-melanoma skin cancer, papillary thyroid cancer, carcinoma in situ of cervical cancer or breast cancer, and localized prostate cancer)
4. Uncontrolled hepatitis B (with the exception of asymptomatic HBsAg-positive or anti-HBcAb-positive cases receiving antiviral prophylaxis such as entecavir or tenofovir)
5. History of chronic hepatitis C (with the exception of HCV IgG positive with a negative HCV-RNA quantification)
6. History of human immunodeficiency virus (HIV) infection
7. Congestive heart failure (NYHA class ≥3)
8. Acute coronary syndrome (new-onset unstable angina or myocardial infarction) or ventricular tachycardia within 6 months prior to study entry
9. History of major neurological or psychiatric illness, including dementia or epilepsy
10. Severe chronic obstructive pulmonary disease with hypoxemia
11. Cerebrovascular disease within 3 months prior to study entry (including transient cerebral ischemia)
12. Unresolved wounds, ulcers, or bone fractures
13. Uncontrolled active infections (viral, bacterial, or fungal infections)
14. Concurrent use of other experimental drugs under investigation
15. Known hypersensitivity to the investigational drugs
16. History of major surgery or serious trauma within 21 days prior to study treatment. Open biopsy within 7 days prior to study treatment
17. Male subjects who had not undergone a vasectomy and have a partner who plans to become pregnant or are unable to use a medically acceptable method of contraception (partner's sterilization or intrauterine device placement, or barrier method combined with diaphragm or condom) during the subject's participation in the study
18. Pregnant or breastfeeding women or women of childbearing potential and men who are not willing to use appropriate methods of contraception during the study
19. Previously treated for T-cell lymphoma with immunotherapy or chemotherapy, except for short-term corticosteroids (for less than 8 days) prior to selection
20. Prior radiotherapy, except for those localized to a single lymph node
21. Central nervous system involvement
22. Contraindication to any of the drugs included in the chemotherapy
23. History of administration of doxorubicin at >200 mg/m²

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response rate | Up to 72 months

SECONDARY OUTCOMES:
overall response rate | Up to 72 months
overall survival | Up to 72 months.
  The time until defined by date of all-cause mortality from the date of IP Administration.
Adverse events | from the day 1 of the clinical trial to 28 days after last drug administration
progression-free survival | Up to 72 months.
  The time until defined by date of all-cause mortality from the date of Investigational Product Administration.
event-free survival | Up to 72 months.
  As the period from enrollment to disease progression/recurrence, treatment for other lymphomas, or death.

OTHER OUTCOMES:
Predictive biomarkers study | Up to 72 months.
  analysis of blood sampling before and after the clinical trial
establishment of treatment response prediction model | Up to 72 months.
  genomic analysis of tumor tissue at diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- 81, Irwon-ro, Gangnam-gu, Seoul, Republic of Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No